CLINICAL TRIAL: NCT00722007
Title: Cormet Hip Resurfacing System Post-PMA Study Group (New Enrollment)
Brief Title: Cormet Post-PMA Study: New Enrollment
Acronym: PASNew
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cormet (P050016) New Enroll
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis
Keywords: hip resurfacing; osteoarthritis; avascular necrosis; rheumatoid arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cormet Hip Resurfacing Post-PMA Group (Experimental): hip resurfacing
  Interventions: Device: Cormet Hip Resurfacing

INTERVENTIONS:
Device: Cormet Hip Resurfacing — Cormet Hip Resurfacing implant
  Other Names: Corin Cormet

SUMMARY:
The primary objective of this study is to evaluate the performance of the Cormet Hip Resurfacing implant system in the post-approval environment.

DETAILED DESCRIPTION:
This study tracks the performance of the Cormet Hip Resurfacing system in the post-approval environment to see if there are significant changes in device performance from the pre-market IDE setting as compared to the post-approval setting. Specifically this study will compare the proportion of subjects achieving a Month 24 composite clinical success (CCS) criterion and 24 month cumulative revision rate among the newly enrolled post-approval study subjects to the IDE subjects' performance on CCS as reported in the Pre-Market Application (PMA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient who meets eligibility criteria consistent with product labeling
* skeletally mature
* mentally capable of completing follow-up forms
* Will be available for follow-up out to 2 years and annually thereafter until the last patient reaches the two-year evaluation
* Has been deemed a candidate for hip replacement by diagnosis of the investigator
* consented to participate in the clinical study

Exclusion Criteria:

* Patient with active or suspected infection in or around the hip joint;
* Patient with bone stock inadequate to support the device
* Patient with severe osteopenia
* Patient with a family history of severe osteoporosis or severe osteopenia;
* Patient with osteonecrosis or avascular necrosis (AVN) with >50% involvement of the femoral head (regardless of FICAT Grade)
* Patient with multiple cysts of the femoral head (>1cm)
* In cases of questionable bone stock, a DEXA scan may be necessary to assess inadequate bone stock.
* Patient with any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery;
* Female of child-bearing age due to unknown effects on the fetus of metal ion release.
* Patient with known moderate or severe renal insufficiency;
* Patient who is immunosuppressed with diseases such as AIDS or person receiving high doses of corticosteroids;
* Patient who is severely overweight;
* Patient with known or suspected metal sensitivity (e.g., jewelry).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2014-04-11 (Actual); Study Completion 2014-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - George Washington University, Washington D.C., District of Columbia
  - Florida Orthopaedic Institute, Tampa, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Lattimore Orthopaedics P.C., Rochester, New York
  - Willamette Orthopedic Group LLC, Salem, Oregon
  - Memorial Bone and Joint Clinic, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 24 Apr 2008 and 21 Dec 2011, 147 participants were enrolled in 6 study hospitals, with 160 Cormet resurfacing implants in 134 unilateral and 13 bilateral procedures.
Units Other Than Participants: Implants
Groups:
- Post-PMA Study: Implanted with Cormet Hip Resurfacing System after pre-market approval.
Period: Overall Study
Arm/Group | Post-PMA Study
Started | 147; 160 Implants
Completed | 117; 128 Implants
Not Completed | 30; 32 Implants

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Groups:
- Cormet Hip Resurfacing Post-PMA Group: Cormet Resurfacing Hip System implanted after pre-market approval
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 147
Number analyzed (Implants) | 160
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [32 to 65]
Sex: Female, Male [Count of Units; unit: Implants]
  Female | 13
  Male | 147
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: The Number of Unilateral Procedures Which Achieved Composite Clinical Success (CCS) at Month 24
Description: Composite Clinical Success (CCS) is based upon the following:
  There has been no revision, removal, or replacement of any device component on or prior to the exact 24 month anniversary (i.e., relative day 730); and Month 24 Harris Hip Total score (HHS) ≥ 80 points.
Time Frame: Month 24+
Measure: Number; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 134
Number analyzed (Implants) | 134
Implants | 104

2. Secondary Outcome: Number of Implants (Unilateral & Bilateral) With Harris Hip Scores (HHS) Components Including Total, Pain & Function Scored at Month 24+
Description: All unilateral and bilateral implants have been assessed using the following grading:
  Total HHS: Excellent (90-100); Good (80-89); Fair (70-79); Poor (<70) Pain HHS: None; Slight; Mild; Moderate; Marked; Totally Disabled Function HHS: Normal (40-47); Mild Dysfunction (30=<39); Moderate Dysfunction (20=<29); Severe Dysfunction (10=<19); Disabled (0=<9)
Time Frame: Month 24+
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 117
Number analyzed (Implants) | 128
Implants
  Total HHS Excellent (90-100) | 109
  Total HHS Good (80-89) | 10
  Total HHS Fair (70-79) | 6
  Total HHS Poor (<70) | 1
  Total HHS missing | 2
  Pain HHS None | 87
  Pain HHS Slight | 28
  Pain HHS Mild | 8
  Pain HHS Moderate | 4
  Pain HHS Marked | 0
  Pain HHS Totally Disabled | 0
  Pain HHS missing | 1
  Function HHS Normal (40-47) | 127
  Function HHS Mild Dysfunction (30=<39) | 1
  Function HHS Moderate Dysfunction (20=<29) | 0
  Function HHS Severe Dysfunction (10=<19) | 0
  Function HHS Disabled (0=<9) | 0

3. Secondary Outcome: Survival Rate Using Kaplan-Meier Survival Curves
Description: Kaplan-Meier survival curves were completed for all implants (unilateral & bilateral) for Month 24
Time Frame: Month 24+
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 147
Number analyzed (Implants) | 160
Implants | 155

4. Secondary Outcome: Number of Procedures (Unilateral & Bilateral) With Any Device Related Adverse Events
Time Frame: Month 24+
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 147
Number analyzed (Implants) | 160
Implants | 9

5. Secondary Outcome: The Number of Procedures (Unilateral & Bilateral) With Any Radiographic Findings at Month 24 Post Operatively
Description: The following was assessed:
  Radiolucency Acetabular Component: I; II; III Radiolucency Femoral Component: Superior; Tip; Inferior Cup Migration and Tilt: Superior/Inferior Migration > 4mm; Medial/Lateral Migration > 4mm; Varus/Valgus Tilt > 4 degrees Stem Migration and Tilt: Subsidence of Femoral Component > 4mm and Stem tilting > 4 degrees Other Assessments: Anteversion of the Head ≥ 5mm; Retroversion of the Head ≥ 5 mm; Hypertrophy in Any Zone; Resorption in Any Zone; Lysis in Any Zone; Osteolysis
Time Frame: Month 24+
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
Number analyzed (Participants) | 115
Number analyzed (Implants) | 126
Implants
  Radiolucency Acetabular Component - I | 1
  Radiolucency Acetabular Component - II | 1
  Radiolucency Acetabular Component - III | 1
  Radiolucency Femoral Component - Superior | 0
  Radiolucency Femoral Component - Tip | 0
  Radiolucency Femoral Component - Inferior | 0
  Superior/Inferior Cup Migration > 4mm | 0
  Medial/Lateral Cup Migration > 4mm | 0
  Varus/Valgus Cup Tilt > 4 degrees | 0
  Stem subsidence of > 4mm and stem tilt of > 4° | 0
  Anteversion of the Head ≥ 5mm | 0
  Retroversion of the Head ≥ 5 mm | 0
  Hypertrophy in Any Zone | 0
  Resorption in Any Zone | 0
  Lysis in Any Zone | 0
  Osteolysis | 0

ADVERSE EVENTS:
Arm/Group | Cormet Hip Resurfacing Post-PMA Group
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 33/147
Other Adverse Events (participants affected / at risk) | 20/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cormet Hip Resurfacing Post-PMA Group (N=147)
Heart valve replacement (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Deep joint infection (Infections and infestations) | 2
Meniscus tear (Injury, poisoning and procedural complications) | 1
Hip pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acetabular loosening (Surgical and medical procedures) | 1
Contralateral hip resurfacing (Surgical and medical procedures) | 15
Contralateral revision THR (Surgical and medical procedures) | 3
Contralateral revision TKR (Surgical and medical procedures) | 1
Contralateral THR (Surgical and medical procedures) | 6
Contralateral TKA (Surgical and medical procedures) | 1
Femoral loosening (Surgical and medical procedures) | 1
Femoral neck fracture (Surgical and medical procedures) | 5
Hip dislocation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cormet Hip Resurfacing Post-PMA Group (N=147)
Hypertension (Cardiac disorders) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Hamstring detachment (Injury, poisoning and procedural complications) | 1
Hip pain (operative side) (Injury, poisoning and procedural complications) | 2
Meniscus tear (Injury, poisoning and procedural complications) | 1
Contralateral hip pain (Musculoskeletal and connective tissue disorders) | 2
Contralateral OA (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Hip pain (operative side) (Musculoskeletal and connective tissue disorders) | 4
Iliopsoas tendonitis (Musculoskeletal and connective tissue disorders) | 1
IT band friction syndrome (Musculoskeletal and connective tissue disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 4
L5-S1 spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Hip dislocation (Surgical and medical procedures) | 1
DVT (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will review publications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. If the sponsor determines the publication contains patentable subject matter the embargo can be extended up to 120 days from the time submitted to the sponsor for review. The PI shall agree to accept the sponsor's reasonable comments and suggestions with respect to publications.